CLINICAL TRIAL: NCT02159560
Title: Uniport and Multiport Epidural Catheters in Post-surgical Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Phillip Hess, Chief of Obstetric Anesthesia, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2014P000085
Record Dates: First submitted 2014-05-19; First posted 2014-06-10 (Estimated); Results first posted 2025-10-29 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Post-operative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Randomized, double-blinded comparison of two epidural catheter designs
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: patient, evaluator, statistician all blinded to assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- End holed catheter (Active Comparator): Single holed, end holed epidural catheter
  Interventions: Device: Epidural catheter
- Three holed catheter (Active Comparator): closed ended, three side holed epidural catheter
  Interventions: Device: Epidural catheter

INTERVENTIONS:
Device: Epidural catheter — The intervention is the use of an end-holed epidural catheter or three-holed side port epidural catheter

SUMMARY:
The investigators hypothesize that multi-port thoracic epidural catheters will provide superior pain relief when compared to uniport catheters for post-surgical patients.

DETAILED DESCRIPTION:
Epidural analgesia (pain relief) is an effective treatment for post-surgical acute pain. The factors that determine the effectiveness of pain relief with epidural analgesia have been studied almost exclusively in the lumbar (low back) spaces for obstetrics (childbirth). These factors include the design of the epidural catheter, the type and dose of medications, and the volume of solution used. One of the important issues specific to the catheter design is whether the tip has a one end-hole, or multiple side holes. The number of holes has been suggested to affect the spread of epidural anesthetic over time, especially with low volume solutions. This has been demonstrated in older, stiffer epidural catheter designs, but has not been shown to be true with the newer, flexible epidural catheters.

The thoracic (upper back) epidural analgesia is widely employed for a many types of surgical pain. While the mechanism of pain relief is similar to that in the lumbar space, there may be differences between the two sites. Firstly, thoracic catheters tend to use low volume, high concentration medication solutions, which likely do not spread as effectively. Secondly, the thoracic catheters often need to be used for prolonged periods of time. Whereas the typical obstetric epidural is used for less than 12 hours, the post-surgical catheter is typically required for one to three days (or more). Finally, the thoracic space is narrow, with a thinner thecal sac, which might promote a difference in the spread of epidural solution.

Thoracic epidural analgesia is routinely used to control post-operative pain for a wide variety of surgical procedures. Based on the improved effectiveness of the one end-hole flexible epidural catheter in obstetrics, this design is commonly used in thoracic epidural analgesia. It has been observed that thoracic epidurals are somewhat less effective after a period of time when compared to the effectiveness of labor epidurals. This may be in part due to the inappropriate assumption that the thoracic epidural space of a post-surgical patient is the same as the lumbar space of a parturient.

The investigators seek to determine whether there is a difference in the analgesia provided by a thoracic multi-port epidural catheter when compared to a thoracic uniport epidural catheter as measured by pain scores, medication given for breakthrough pain, and need to add intravenous opioids. As mentioned previously, these catheters have been studied extensively in laboring patients but there is a striking paucity of literature regarding how anesthetic solutions spread in the thoracic epidural spaces of non-pregnant post-surgical patients and how this may be affected by catheter type. If the hypothesis is supported by results, it may change the practice within the study institution, and possibly, on a much larger scale. This study may also provide a foundation for further research into the physiology of the thoracic epidural space, how it differs from the lumbar epidural space, and how a medication solution spreads within this unique space.

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* Surgery in the thorax or upper abdomen
* Age between 18 and 75
* Expected use of epidural analgesia for >24 hours

Exclusion Criteria:

* Contraindication to epidural catheterization
* Chronic use of opioids
* Chronic pain
* Allergy to the standard medications used
* Body Mass Index >40
* Delirium
* Dementia

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2014-06; Primary Completion 2021-12 (Actual); Study Completion 2021-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philip E Hess, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Enrolled
Arm/Group | End Holed Catheter | Three Holed Catheter
Started | 120 | 120
Completed | 83 | 83
Not Completed | 37 | 37
Period: Analyzed
Arm/Group | End Holed Catheter | Three Holed Catheter
Started | 83 | 83
Completed | 76 | 79
Not Completed | 7 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | End Holed Catheter | Three Holed Catheter | Total
Number analyzed (Participants) | 76 | 79 | 155
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.7 (8.8) | 58.6 (10.4) | 60.3 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 43 | 79
  Male | 40 | 36 | 76
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 8 | 14
  Not Hispanic or Latino | 70 | 71 | 141
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 7 | 10 | 17
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 14 | 17 | 31
  White | 51 | 45 | 96
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 7 | 11

OUTCOME MEASURES:

1. Primary Outcome: Epidural Catheter Failure
Description: The primary outcome of the study will be the incidence of failed epidural analgesia, defined as the need to add intravenous opioids or halting or replacing the epidural catheter because of lack of pain control.
Time Frame: 72 hours
Measure: Count of Participants; unit: Participants
Arm/Group | End Holed Catheter | Three Holed Catheter
Number analyzed (Participants) | 76 | 79
Participants | 52 | 51

2. Secondary Outcome: Number of Subjects Receiving Supplemental Treatments
Description: number of subjects receiving supplemental treatments required to maintain continual comfort
Time Frame: 72 hours
Measure: Count of Participants; unit: Participants
Arm/Group | End Holed Catheter | Three Holed Catheter
Number analyzed (Participants) | 76 | 79
Participants | 30 | 29

3. Other Pre Specified Outcome: Median Dose of Medication
Description: Median dose (per hour) of medication required to maintain comfort
Time Frame: 72 hours
Measure: Median (Inter-Quartile Range); unit: ml per hour
Arm/Group | End Holed Catheter | Three Holed Catheter
Number analyzed (Participants) | 76 | 79
ml per hour | 8 [7 to 10] | 9 [7 to 10]

ADVERSE EVENTS:
Time Frame: 72 hours
Arm/Group | End Holed Catheter | Three Holed Catheter
All-Cause Mortality (participants affected / at risk) | 0/76 | 0/79
Serious Adverse Events (participants affected / at risk) | 0/76 | 0/79
Other Adverse Events (participants affected / at risk) | 0/76 | 0/79

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-02-12): https://cdn.clinicaltrials.gov/large-docs/60/NCT02159560/Prot_SAP_000.pdf